CLINICAL TRIAL: NCT06047535
Title: Naxitamab and Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF) Combined With Isotretinoin for Maintenance Treatment of Patients With High-Risk Neuroblastoma in First Complete Response. A Single-Arm, Multicenter Clinical Trial
Brief Title: Naxitamab and Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF) Combined With Isotretinoin for Maintenance Treatment of Patients With High-Risk Neuroblastoma in First Complete Response.
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: SciClone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ONN203
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Neuroblastoma
Keywords: high-risk neuroblastoma with first complete response
MeSH Terms: conditions — Neuroblastoma | interventions — naxitamab; Granulocyte-Macrophage Colony-Stimulating Factor; Isotretinoin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Naxitamab — Naxitamab + GM-CSF:
  Cycles 1-5: Patients will receive naxitamab IV at 3 mg/kg/infusion on Day 1, 3 and 5 and GM-CSF sc at 5 µg/kg/day on Days -4 to 0 and at 10 µg/kg/day on Days 1-5 for 5 cycles.
  Isotretinoin:
  Cycles 3-8: Patients will receive isotretinoin PO at 160 mg/m2/day divided into two daily doses on Days 15-28 for 6 cycles.
  Other Names: GM-CSF; isotretinoin

SUMMARY:
This is a single-arm, multicenter clinical trial conducted in patients ≥ 12 months of age with high-risk neuroblastoma in first complete response. 62 patients will be enrolled to receive naxitamab + GM-CSF in combination with isotretinoin.

In line with post-consolidation maintenance treatment of high-risk neuroblastoma, this trial will include patients with high-risk neuroblastoma in first complete response. Patients must have completed a multimodal frontline regimen (induction and consolidation) and have achieved complete response (positive bone marrow minimal residual disease as assessed by RTqPCR is allowed) following the multi agent induction and consolidation therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Documented NB at time of diagnosis defined as26:

   1. histopathology of solid tumor biopsy, or
   2. BM aspirate or biopsy indicative of NB plus high blood or urine catecholamine metabolite levels
2. Documented high-risk disease at time of initial diagnosis defined as24, 26:

   1. MYCN-amplified at stage L2, M or MS (according to International Neuroblastoma Risk Group (INRG)) of any age or
   2. MYCN-nonamplified with stage M (according to INRG) and diagnosed at ≥ 18 months of age or
3. Subjects must have completed frontline therapy described in 6.3.2 and have verified complete response according to INRC25 (BM MRD is allowed as assessed by RTqPCR at site28) after completion of induction and consolidation with or without ASCT
4. Age ≥ 12 months at trial enrollment
5. Life expectancy of greater than 6 months, as judged by the Investigator
6. Written informed consent from legal guardian(s) and/or patient in accordance with local regulations. Children must provide assent as required by local regulations

Exclusion Criteria:

1. Verified PD during induction or consolidation therapy
2. Any systemic anti-cancer therapy, including chemotherapy, within 3 weeks prior to enrollment
3. ASCT within 6 weeks prior to enrollment or ongoing toxicity caused by the ASCT at the discretion of the Investigator
4. Therapeutic 131I-MIBG within 6 weeks prior to enrollment
5. Prior anti-GD2 therapy
6. Performance status of < 50% as per the Lansky scale (patients less than 16 years of age) or Karnofsky scale (patients aged 16 years or older)
7. Left ventricular ejection fraction < 50% by echocardiography
8. Inadequate pulmonary function defined as evidence of dyspnea at rest, exercise intolerance, and/or chronic oxygen requirement. In addition, room air pulse oximetry < 94% and/or abnormal pulmonary function tests if these assessments are necessary at the discretion of the Investigator
9. Life threatening infection(s)
10. Treatment with long-acting myeloid growth factor within 14 days or short-acting myeloid growth factor within 7 days prior to first dose of GM-CSF
11. Treatment with immunosuppressive agents (local steroids excluded) within 4 weeks prior to enrollment
12. History of allergy or known hypersensitivity to GM-CSF, E. coli-derived products, or any component of GM-CSF, naxitamab, isotretinoin or vitamin A.
13. NB in the Central Nervous System (CNS) or leptomeningeal disease within 6 months prior to enrollment
14. Patients with uncontrolled seizure disorders despite anticonvulsant therapy (defined as a seizure event within 3 months prior to enrollment)
15. Unacceptable hematological status prior to first dosing, defined as one of the following:

    1. Hemoglobin <5.0 mmol/L (<8 g/dL)
    2. White blood cell (WBC) count <1000/µL
    3. Absolute neutrophil count (ANC)<750/µL
    4. Platelet count <75,000/µL
16. Unacceptable liver function prior to first dosing, defined as one of the following:

    1. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) >5 times upper normal limit (UNL)
    2. Bilirubin >1.5 x UNL
17. Unacceptable kidney function prior to first dosing, defined as:

    a. Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2 calculated by the 2009 revised Bedside Schwartz Equation27 (Please refer to Appendix 1)
18. Inability to comply with protocol, as judged by the Investigator
19. Patients with a significant intercurrent illness (any ongoing serious medical problem unrelated to cancer or its treatment) that is not covered by the detailed exclusion criteria and that is expected to interfere with the action of trial agents or to significantly increase the severity of the toxicities experienced from trial treatment
20. Females of childbearing potential who are pregnant, breast feeding, intend to become pregnant, or are not using adequate contraceptive methods or males who are not using adequate contraceptive methods. Contraception must be used for 1 month after last isotretinoin treatment and 42 days after last naxitamab treatment whichever comes last for both genders

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-10-31 (Estimated); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-08-15 (Estimated)

PRIMARY OUTCOMES:
2-year progression free survival | 2 years
  2-year progression free survival defined as the proportion of patients alive and without progressive disease or relapse 2 years after enrollment